CLINICAL TRIAL: NCT03581825
Title: Clinical Evaluation of a Reusable Multifocal Optical Design in a Presbyopic Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6201
Record Dates: First submitted 2018-06-26; First posted 2018-07-10 (Actual); Results first posted 2020-04-29 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Myopic subjects who are habitual soft contact lens wearers between the ages of 40 and 70 years of age, will be randomized to sequence Test/Control. Alternative Spherical lenses will be used if optimization cannot be achieved with the Multifocal lenses.
  Interventions: Device: senofilcon A Multifocal; Device: senofilcon A Sphere; Device: etafilcon A Multifocal; Device: etafilcon A Sphere
- Control/Test (Experimental): Myopic subjects who are habitual soft contact lens wearers between the ages of 40 and 70 years of age, will be randomized to sequence Control/Test. Alternative Spherical lenses will be used if optimization cannot be achieved with the Multifocal lenses.
  Interventions: Device: senofilcon A Multifocal; Device: senofilcon A Sphere; Device: etafilcon A Multifocal; Device: etafilcon A Sphere

INTERVENTIONS:
Device: senofilcon A Multifocal — JJVC Investigational Multifocal Contact Lens
Device: senofilcon A Sphere — ACUVUE OASYS 2-WEEK with HYDRACLEAR PLUS
Device: etafilcon A Multifocal — 1-Day Acuvue Moist Brand Multifocal Contact Lens
Device: etafilcon A Sphere — 1-Day Acuvue Moist Brand Contact Lens

SUMMARY:
This is a single-masked, randomized-controlled, dispensing clinical trial. A total of approximately 60 eligible myopic subjects will be targeted to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. The subject must be between 40 and 70 years of age (inclusive).
  4. The subject's distance spherical equivalent refraction must be in the range of -1.25 D to -3.75 D in each eye.
  5. The subject's refractive cylinder must be ≤0.75 D in each eye.
  6. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
  7. The subject must have distance best corrected visual acuity of 20/20-3 or better in each eye.
  8. Subjects must own a wearable pair of spectacles if required for their distance vision.
  9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
  10. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

      Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating.
  2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
  3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
  4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
  5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
  6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, cataract surgery, retinal surgery, etc.).
  7. A history of amblyopia, strabismus or binocular vision abnormality.
  8. Any current ocular infection or inflammation.
  9. Any current ocular abnormality that may interfere with contact lens wear.
  10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.
  11. Use of any ocular medication, with the exception of rewetting drops.
  12. History of herpetic keratitis.
  13. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
  14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
  15. Any known hypersensitivity or allergic reaction to Optifree®Replenish® multipurpose care solution or Eye-Cept® rewetting drop solution.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Coughlin Eye Center, Orlando, Florida
  - VisionCare Associates, East Lansing, Michigan
  - Eyecare Management Company, LLC, Raytown, Missouri
  - Jamestown Optometric Group, Jamestown, New York
  - Susquehanna Eye Care, Vestal, New York
  - Bryan Frazier, OD, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 63 subjects were enrolled in this study. Of those, 62 were dispensed at least 1 study lens. Of those dispensed a study lens, 60 subjects completed the study while 2 were discontinued from the study.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the Control lens during the second period
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 31 | 31
Completed | 30 | 31
Not Completed | 1 | 0
Not completed — Lens Discomfort | 1 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 30 | 31
Completed | 30 | 30
Not Completed | 0 | 1
Not completed — Unsatisfactory Vision to Test | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: All subjects dispensed a study lens
Arm/Group | Total
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (6.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 12
Race/Ethnicity, Customized [Number; unit: Participants]
  Black or African American | 3
  White | 59
Region of Enrollment [Number; unit: Participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: CLUE Vision
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 2-Week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test: Subjects that wore the Test lens in either the first or second period of the study.
Arm/Group | Test
Number analyzed (Participants) | 53
units on a scale | 57.1 (19.16)
Statistical Analysis 1: Comparison: Test; Test type: Superiority — Statistically superiority was concluded if the lower limit of the confidence intervals of the Test lens are greater than 40 points; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean = 56.3, 95% CI 2-sided [51.2 to 61.4], Standard Error of Mean 2.55

2. Secondary Outcome: CLUE Vision Comparison Between Test and Control
Description: as for outcome 1
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Test | Control
Number analyzed (Participants) | 53 | 53
units on a scale | 57.1 (19.16) | 53.3 (18.55)
Statistical Analysis 1: Comparison: Test vs Control; Test type: Non-Inferiority — The non-inferiority of the Test lens relative to the Control was concluded if the lower confidence limit of LSM difference was above the non-inferiority margin -5; Linear Mixed Model; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = 3.4, 95% CI 2-sided [-0.5 to 7.4], Standard Error of Mean 2.00 — Mean Difference was calculated as Test minus Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 5 weeks per subject.
Arm/Group | Test | Control
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/62
Other Adverse Events (participants affected / at risk) | 0/62 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT03581825/Prot_SAP_000.pdf